CLINICAL TRIAL: NCT06021756
Title: A Single-center Phase I Open-label Study of the Tolerability and Efficacy of Low-dose Ketamine Infusion for Treatment of Levodopa-Induced Dyskinesia in Patients With Parkinson's Disease
Brief Title: Phase I Open-label Study of Low-dose Ketamine Infusion Treatment in Levodopa-Induced Dyskinesia in Parkinson's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arizona (Other)
Collaborators: Scott Richards (Unknown)
Responsible Party: Principal Investigator, Scott Sherman, Scott J. Sherman MD, PhD,, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1903472458_ MOD00004091
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Levodopa-Induced Dyskinesia; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention: Ketamine (Experimental): Ketamine will be administered as intravenous infusions with infusion rates ranging from 0.05 mg/kg/hr to 0.30 mg/kg/hr.
  Interventions: Drug: Intervention: Ketamine

INTERVENTIONS:
Drug: Intervention: Ketamine — Ketamine will be administered as intravenous infusions with infusion rates ranging from 0.05 mg/kg/hr to 0.30 mg/kg/hr.
  Other Names: Intervention: Ketamine i.v.

SUMMARY:
The primary objective is to determine the tolerability and efficacy of a low-dose ketamine infusion for the treatment of Levodopa-Induced dyskinesias (LID), both acutely and during post-infusion evaluation (week 2-6), as measured by a change in patient diaries of dyskinesia and the UDysRS. Secondary objectives include observing the effects of ketamine on various symptoms of Parkinson's disease and Levodopa side effects. This includes the duration of "off," "on without dyskinesia," and "troublesome dyskinesia" time during waking hours, effects on chronic and acute pain, quality of life, and other general PD symptoms as noted in the Unified Parkinson's Disease Rating Scale.

There is no highly effective treatment for levodopa-induced dyskinesia. This research study will use intermittent infusions of ketamine, on 10 volunteer subjects, which could provide significant improvement in dyskinesia utilizing a novel mechanism of action compared to current treatment strategies. Positive results in this study could lead to new novel treatments for dyskinesia and further development for other PD symptoms such as depression and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's Disease as defined by the UK Parkinson's Disease Society Brain Bank Criteria
* Be male or female between ages 30-85
* Be on at least two years of treatment of levodopa of at least 400 mg or 4mg/kg daily
* Have levodopa induced dyskinesia for at least 2 hours per day
* Have been on stable doses of all anti-Parkinson's medications for 30 days and be willing to remain on the same doses throughout the course of the study
* The subject/caregiver must demonstrate ability to complete an accurate home diary based on training and evaluation (visit 2)
* Female subjects not of childbearing potential

  * infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenesis; or
  * post-menopausal - defined as either

    * A woman at least 40 years of age with an intact uterus, not on hormone therapy, who has had at least 1 year of spontaneous amenorrhea with a follicle-stimulating hormone level >40 mIU/mL
    * A woman 55 or older not on hormone therapy, who has had at least 6 months of spontaneous amenorrhea
    * A woman at least 55 years of age with a diagnosis of menopause prior to start of hormone replacement therapy.
* Male subjects, regardless of their fertility status, with nonpregnant women of childbearing potential (WOCBP) partners must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use a highly effective (less than 1% failure rate) method of contraception (such as combination oral contraceptives, implanted contraceptives, or intrauterine devices) or effective method of contraception (such as diaphragms with spermicide or cervical sponges) for the duration of the study and until their plasma concentrations are below the level that could result in a relevant potential exposure to a possible fetus, predicted to be 90 days following the last dose of study drug.

  * Men and their partners may choose to use a double-barrier method of contraception. (Barrier protection methods without concomitant use of a spermicide are not an effective or acceptable method of contraception. Thus, each barrier method must include use of a spermicide. It should be noted, however, that the use of male and female condoms as a double barrier method is not considered acceptable due to the high failure rate when these barriers' methods are combined). Men with pregnant partners should use condoms during intercourse for the duration of the study and until the end of estimated relevant potential exposure in WOCBP (90 days).
  * Men should refrain from sperm donation for the duration of the study and until their plasma concentrations are below the level that could result in a relevant potential exposure to a possible fetus, predicted to be 90 days following the last dose of study drug.

Exclusion Criteria:

* Diagnosis of an atypical or secondary parkinsonian syndrome
* Lack of documented response to levodopa
* Prior exposure to ketamine within the last one year
* Significant history of premorbid psychiatric illness other than depression
* Currently taking psychotropic medications with significant dopamine receptor blocking effects such as first-generation antipsychotic agents (clozapine, quetiapine, pimavanserin are allowed as concomitant medications - see section 5.4)
* Have used antipsychotic medications, with the exception of clozapine, quetiapine, pimavanserin in the 6 months prior to screening (Visit 1) and at any time during the course of the study
* Cognitive impairment as demonstrated as a score of 20 or below on the Montreal Cognitive Assessment (MoCA)
* Has a history of drug or alcohol dependence or abuse
* History of visual or auditory hallucinations (visual hallucinations will be acceptable if scored 2 or less on UPDRS II)
* Serious or unstable medical condition that would increase risk in view of the principal investigator.
* The subject is female, and is pregnant or lactating at the time of pregnancy or has positive pregnancy test result at screening.
* Baseline BP >160/95 on average of three readings at the screening visit
* History of arrhythmia, unstable angina, or significant cardiac dysfunction
* Have significant central nervous system disease, other than PD, that may affect cognition or the ability to complete the study, including but not limited to other dementias (e.g., Alzheimer's disease [AD]).
* Have a history in the last 6 months of transient ischemic attacks or stroke.
* Have a history of intracerebral hemorrhage due to hypertension.
* Have a history of hypertensive encephalopathy.
* If the Investigator believes that the subject would not be a good fit for the study for any reason.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Change in the Unified Dyskinesia Rating Scale (UDysRS) total score | 2 and 12 weeks
  Change in the Unified Dyskinesia Rating Scale (UDysRS) total score from Baseline to Week 2 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Sherman, Principal Investigator — University of Arizona Health Sciences Center - Dep. of Neurology
Locations (1):
- Scott J Sherman, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No